CLINICAL TRIAL: NCT04328090
Title: Evaluation of the Potential Impact of Computerized Antimicrobial Stewardship on the Antimicrobial Use After Cardiovascular Surgeries
Brief Title: Evaluation of the Potential Impact of Computerized Antimicrobial Stewardship
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Shengshou Hu, Professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-ZX10
Record Dates: First submitted 2020-03-17; First posted 2020-03-31 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Antimicrobial Stewardship; Cardiovascular Surgeries; Computerized Decision Support System; Coronary Artery Disease; Valve Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDSS-Antimicrobial stewardship (Experimental): Computer-based, multicomponent intervention targeting on reduction of perioperative antimicrobial use will be delivered to teams in the intervention arm.
  Interventions: Other: Computer based Antimicrobial stewardship (AMS) intervention system
- Standard of care (No Intervention): Teams in the control arm will continue with usual standard clinical care.

INTERVENTIONS:
Other: Computer based Antimicrobial stewardship (AMS) intervention system — 1. Re-evaluation alerts and decision support for the duration of antimicrobial treatment.
  2. Re-evaluation alerts and decision support for the choice of antimicrobial.
  3. Quality control audit and feedback.
  Arms: CDSS-Antimicrobial stewardship

SUMMARY:
This trial is an open-label, two-arm, cluster-randomized, controlled trial with cardiovascular surgical teams as the unit of randomization. Eligible teams with written consent are randomized to the intervention or control arm by random number generator. Computer-based, multicomponent intervention targeting on reduction of perioperative antimicrobial use will be delivered to teams in the intervention arm. Teams in the control arm will continue with usual clinical care.

DETAILED DESCRIPTION:
The aim of the EPIC trial is to assess if a multicomponent computer-based system incorporated into the workflow can reduce days of therapy (DOT) per admission after cardiovascular surgeries in the intervention surgical teams compared with controlled surgical teams, over a one-year period. This trial is an open-label, two-arm, cluster-randomized, controlled trial with cardiovascular surgical teams as the unit of randomization. Eligible teams with written consent are randomized to the intervention or control arm by random number generator. Computer-based, multicomponent intervention targeting on reduction of perioperative antimicrobial use will be delivered to teams in the intervention arm. Teams in the control arm will continue with usual clinical care. The intervention includes re-evaluation alerts and decision support for the duration of antimicrobial treatment, re-evaluation alerts and decision support for the choice of antimicrobial, and quality control audit and feedback. Nine teams per arm with an average size of 1125 admissions will be recruited. Primary outcome will be the overall systemic antibiotic use measured in DOT of systemic antibiotic use per admission. Secondary outcomes include a series of indices to evaluate antimicrobial use, microbial resistance, perioperative infection outcomes, patient safety, resource consumption and user compliance/satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age;
2. Receiving at least one open-chest cardiovascular surgery during the same admission.

Exclusion Criteria:

1. Intravenous or oral antimicrobial use within two weeks before surgery;
2. Emergent/urgent surgery;
3. Admitted for isolated stenting or heart transplantation or implantation of ventricular assist device or implantation of extracorporeal membrane oxygenation;
4. Admitted for subacute bacterial endocarditis;
5. Length of ICU stay over 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2473 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Days of antimicrobial therapy (DOT) per admission | From the date of admission to the date of discharge, assessed up to 3 months.
  DOT represents a specific antibiotic administered to an individual patient on a calendar day independent of dose and route.
DOT per 1000 patient-days (PD) | From the date of admission to the date of discharge, assessed up to 60 days.
  DOT per 1000 patient-days

SECONDARY OUTCOMES:
Drug usage (DDDs) per 100 PD | From the date of admission to the date of discharge, assessed up to 60 days.
  Items issued × Amount of drug per item per 100 PD
Drug usage (DDDs) per admission | From the date of admission to the date of discharge, assessed up to 60 days.
  Items issued × Amount of drug per item per admission
Length of therapy (LOT) per 100 PD | From the date of admission to the date of discharge, assessed up to 60 days.
  Number of days during which antimicrobial is used per 100 PD
Length of therapy (LOT) per admission | From the date of admission to the date of discharge, assessed up to 60 days.
  Number of days during which antimicrobial is used per admission
Days per treatment period overall and for specific indications | From the date of admission to the date of discharge, assessed up to 60 days.
  treatment period: antibiotic treatment not interrupted by more than one calendar day or discharge.
Rate of participants with clostridium difficile colitis | From the date of admission to the date of discharge, assessed up to 60 days.
  Colitis associated with Clostridium difﬁcile infection
Incident clinical cultures with multidrug resistant organisms (MRSA, ESBL-E, CRE, VRE, or Pseudomonas aeruginosa) per 1000 PD and admission. | From the date of admission to the date of discharge, assessed up to 60 days.
  MRSA=methicillin-resistant Staphylococcus aureus; ESBL-E=extended spectrum beta-lactamase producing Enterobacteriaceae; CRE=Carbapenem resistant Enterobacteriaceae; VRE=vancomycin-resistant enterococci.
In-hospital or 30-day surgical site infections (SSIs) | 30 days from accomplished of the surgery.
  Occurs within 30 days postoperatively and involves skin or subcutaneous tissue of the incision and at least one of the following: (1) purulent drainage from the incision, (2) organisms isolated from an aseptically obtained culture of fluid or tissue from the incision, (3) at least one of the following signs or symptoms of infection: pain or tenderness, localized swelling, redness, or heat, and incision is deliberately opened by surgeon and is culture-positive or not cultured (a culture-negative finding does not meet this criterion), and (4) diagnosis of SSI by the surgeon or attending physician.
Rate of in-hospital bloodstream infections | From the date of admission to the date of discharge, assessed up to 60 days.
  Blood stream infection after surgery (ICD 10: A41.9)
Rate of in-hospital pneumonia | From the date of admission to the date of discharge, assessed up to 60 days.
  Pulmonary infection after surgery (ICD 10：J98.402)
In-hospital or 30-day mortality, postoperative | 30 days from accomplished of the surgery or within hospital.
  mortality with in 30-day after the surgery
In-hospital or 30-day myocardial infarction (MI), postoperative and newly onset | 30 days from accomplished of the surgery or within hospital.
  MI (in accordance with the fourth edition of MI definition) was termed type 5 MI, procedure related MI. Briefly, the criteria are as follows:
  1. Elevation of cardiac troponin (cTn)>10 times of the 9th percentile upper reference limit with patients with normal baseline;
  2. For patients with elevated preprocedural cTn values, elevation of cTn>10 fold increase and manifest a change from the baseline value of over 20%;
  3. With as least one of the following:
  4. Development of new pathological Q waves;
  5. Imaging evidence of loss of viable myocardium that is presumed to be new and in a pattern consistent with an ischemic aetiology;
  6. Angiographic findings consistent with a procedural flow-limiting complication.
In-hospital or 30-day stroke, postoperative and newly onset | 30 days from accomplished of the surgery or within hospital
  Stroke refers to newly onset stroke after surgery (ICD 10: I60.0-I60.9; I61.0-I61.9; I62.0; I62.1; I62.9; I63.0-I63.9; I64)
In-hospital or 30-day acute kidney injury (AKI) , postoperative and newly onset | 30 days from accomplished of the surgery or within hospital
  AKI refers to newly onset AKI after surgery
  1. Acute renal dysfunction within 48 hours (ICD 10: N17);
  2. AKI stage I: creatinine≥26.5µmol/L; creatinine over 1.5-1.9 times of baseline value; urine output<0.5ml/kg/hour for 6-12
Length of hospital stay (LOS) | From the date of admission to the date of discharge, assessed up to 60 days.
  Length of hospital stay (LOS)
Costs of administered antimicrobials (overall and by class) per admission | From the date of admission to the date of discharge, assessed up to 60 days.
  Costs of administered antimicrobials (overall and by class) per admission
Total costs of hospitalization | From the date of admission to the date of discharge, assessed up to 60 days.
  Total costs of hospitalization
User satisfaction with the system | From the date of inclusion of the first patient to the date of discharge of the last patient, assessed up to 12 months.
  Using questionnaire and an interview guide for the process evaluation of the intervention system.
User compliance with the system | From the date of inclusion of the first patient to the date of discharge of the last patient, assessed up to 12 months.
  Ccompliance with the multicomponent intervention protocols will be assessed. This will be done by evaluating the total number of times the intervention tools fail to change the physicians' decision on antimicrobial prescription over the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Xin Yuan, PhD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital; Kai Chen, PhD, Study Director — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuan X, Chen K, Yuan J, Chu Q, Hu S, Gao Y, Yu F, Diao X, Chen X, Li Y, Sun H, Shu C, Wang W, Pan X, Zhao W, Hu S. Evaluation of the effectiveness and safety of a multi-faceted computerized antimicrobial stewardship intervention in surgical settings: A single-centre cluster-randomized controlled trial. Int J Antimicrob Agents. 2023 May;61(5):106787. doi: 10.1016/j.ijantimicag.2023.106787. Epub 2023 Mar 17. PMID 36935089
- [Derived] Yuan X, Chen K, Zhao W, Hu S, Yu F, Diao X, Chen X, Hu S. Open-label, single-centre, cluster-randomised controlled trial to Evaluate the Potential Impact of Computerisedantimicrobial stewardship (EPIC) on the antimicrobial use after cardiovascular surgeries: EPIC trial study original protocol. BMJ Open. 2020 Nov 26;10(11):e039717. doi: 10.1136/bmjopen-2020-039717. PMID 33243799